CLINICAL TRIAL: NCT06029673
Title: Cabergoline for Lactation Inhibition After Early Second-Trimester Abortion or Pregnancy Loss: A Randomized Controlled Trial
Brief Title: Cabergoline for Lactation Inhibition After Early Second-Trimester Abortion or Pregnancy Loss
Acronym: eLISTA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Planned Parenthood Mar Monte (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 71540
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Results first posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Lactation Suppressed
Keywords: abortion; fetal demise; lactation; engorgement
MeSH Terms: conditions — Fetal Death; Breast Feeding; Hyperemia | interventions — Cabergoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cabergoline (Experimental): After the completion of the surgical procedure or medical induction for the early second-trimester abortion or fetal loss, the participant will be administered cabergoline 1mg orally with juice or water by the clinician or study investigator.
  Interventions: Drug: Cabergoline 1 MG
- Placebo (Placebo Comparator): After the completion of the surgical procedure or medical induction for the early second-trimester abortion or fetal loss, the participant will be administered a placebo pill orally with juice or water by the clinician or study investigator.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cabergoline 1 MG — Dopamine agonist
  Other Names: Dosintex
  Arms: Cabergoline
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Breast pain following second-trimester abortion is common. Breast engorgement and milk leakage following second-trimester perinatal loss and abortion can cause both physical pain and emotional distress. Dopamine agonists have previously been shown to be effective in lactation inhibition for third-trimester fetal/neonatal loss or contraindications to breastfeeding. The investigator's prior work demonstrated that compared to placebo, a single dose of cabergoline was effective in preventing breast symptoms after abortion or loss 18-28 weeks. As lactogenesis starts as early as 16 weeks gestation, the investigators hope to determine the efficacy of cabergoline earlier in the second trimester,16-20 weeks.

DETAILED DESCRIPTION:
This study is a double-blinded, placebo-controlled, gestational-age stratified superiority trial of those undergoing abortion or intrauterine fetal demise between 16 and 20-weeks gestation at Stanford Health Care. Participants will be randomized to either cabergoline 1 mg or placebo the day of procedure. Participants will complete a survey to assess symptoms, using the validated Bristol Breast Symptoms Inventory, and side-effects at baseline and Day 2, 4, 7, and 14 after the procedure. The study plan is to recruit 72 subjects powered to detect a 45% decrease in those reporting breast symptoms compared to the control group.

This study has the potential to improve overall patient experience by validating the routine use of cabergoline for lactation inhibition in the early second-trimester after abortion or pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant people, ages 18 years or older
* Intrauterine pregnancy between 16/0-19/6 weeks of gestation age (by ultrasound dating performed prior to or same day of enrollment visit)
* Consented for an induced, elective abortion or undergoing management of fetal demise
* English or Spanish speaking
* Able to consent for a research study, literate in English or Spanish
* Willing to comply with study procedures and follow-up
* Access to smart phone throughout study

Exclusion Criteria:

18 Years Female No No

Inclusion Criteria:

* Pregnant people, ages 18 years or older
* Intrauterine pregnancy between 18/0-28/0 weeks of gestation age (by ultrasound dating performed prior to or same day of enrollment visit)
* Consented for an induced, elective abortion or undergoing induction for demise
* English or Spanish speaking
* Able to consent for a research study, literate in English or Spanish
* Willing to comply with study procedures and follow-up
* Access to smart phone throughout study

Exclusion Criteria:

* Prior mastectomy (breast reduction or chest masculinization surgery acceptable)
* Currently breastfeeding
* Currently receiving dopamine agonist or antagonist therapy for other indication leg syndrome)
* Contraindication to cabergoline (as per package insert)
* Uncontrolled hypertension - defined as baseline BP > 160/110, or chronic hypertension requiring more than one baseline medication, or current pregnancy-induced hypertension spectrum disorders (gestational hypertension, preeclampsia, eclampsia)
* History of cardiac valvular disorders or valvular repair
* History of pulmonary, pericardial, or retroperitoneal fibrotic disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Planned Parenthood - San Jose Central Health Center, San Jose, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be requested for meta-analysis inclusion
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Henkel A, Cahill EP, Chavez S, Shorter JM, Amaya SI, Kaur S, Soltani A, Caron J, Crowe S, Williams Z, Mastey N, Lyell DJ, Shaw KA. Cabergoline for Lactation Inhibition After Early Second-Trimester Abortion or Pregnancy Loss: A Randomized Controlled Trial. Obstet Gynecol. 2026 Feb 1;147(2):277-284. doi: 10.1097/AOG.0000000000006137. Epub 2025 Dec 5. PMID 41538804

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabergoline: After the completion of the surgical procedure or medical induction for the early second-trimester abortion or fetal loss, the participant is administered cabergoline 1mg orally with juice or water by the clinician or study investigator.
- Placebo: After the completion of the surgical procedure or medical induction for the early second-trimester abortion or fetal loss, the participant is administered a placebo pill orally with juice or water by the clinician or study investigator.
Period: Overall Study
Arm/Group | Cabergoline | Placebo
Started | 34 | 35
Completed | 32 | 34
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis - participants that did not provide any additional surveys beyond date of enrollment were excluded
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabergoline | Placebo | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 32 | 34 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (7.9) | 28.6 (7.2) | 28.2 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 34 | 66
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 7 | 18 | 25
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 18 | 6 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 34 | 66
Prior breastfeeding experience [Count of Participants; unit: Participants] | 11 | 17 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Breast Pain
Description: Participants will assess their breast symptoms using the validated Bristol Breast Inventory survey to assess 4 domains of breast symptoms: tenderness, engorgement, leaking milk, pain relief. Participants who indicated symptoms in any of these areas met the criteria for this outcome.
Time Frame: Day 4 after procedure
Population: ITT analysis - participants that did not provide any additional surveys beyond date of enrollment were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 32 | 34
Participants | 16 | 30

2. Secondary Outcome: Number of Participants Experiencing Side-effects
Description: Participants selected from previously documented side-effects from the dopaminergic class or entered as free-text. Participants may have reported more than one side-effect. The experience of dopaminergetic medication side effects may or may not be considered to be adverse events.
Time Frame: Cumulative over 2 weeks
Population: ITT analysis - participants that did not provide any additional surveys beyond date of enrollment were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 32 | 34
Participants | 26 | 31

3. Secondary Outcome: Number of Participants Reporting Significant Bother From Breast Pain
Description: Assessed using a Facial Pain Score; scale range 0-6 (higher scores indicate greater pain), with significant bother >=4
Time Frame: Day 4 after procedure
Population: ITT analysis - participants that did not provide any additional surveys beyond date of enrollment were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 32 | 34
Participants | 1 | 7

4. Secondary Outcome: Number of Participants Reporting Significant Bother From Side-effects
Description: Assessed using a Facial Pain Score; scale range 0-6 (higher scores indicate greater pain), with significant bother >=4
Time Frame: Cumulative over 2 weeks
Population: ITT analysis - participants that did not provide any additional surveys beyond date of enrollment were excluded
Measure: Count of Participants; unit: Participants
Arm/Group | Cabergoline | Placebo
Number analyzed (Participants) | 32 | 34
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: 14 days following drug/placebo allocation
Arm/Group | Cabergoline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT06029673/Prot_SAP_000.pdf